CLINICAL TRIAL: NCT03117842
Title: Using a Theory-based SMS/VM Intervention to Improve Sexual and Reproductive Health of Female Entertainment Workers in Cambodia: Study Protocol of a Randomized Controlled Trial
Brief Title: Using a Theory-based SMS/VM Intervention to Improve Sexual and Reproductive Health of Female Entertainment Workers in Cambodia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Touro University, California (Other)
Collaborators: KHANA Center for Population Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: mobilelinkcambodia
Record Dates: First submitted 2017-03-31; First posted 2017-04-18 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Reproductive Health; Sexual Health
Keywords: Female entertainment workers; mHealth; HIV testing; Cambodia

STUDY DESIGN:
Intervention Model Description: A 12-month randomized controlled trial (RCT) will be conducted to evaluate the Mobile Link intervention, with two arms of 300 FEWs each. FEWs will be equally randomized into one of two groups: (1) no intervention and (2) SMS or VM theory-based behavioral messages.
Who Masked: Outcomes Assessor
Masking Description: Statistical Analysis will be conducted without knowledge of the assignment of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will receive the 3 text or voice messages weekly. The messages will be designed to enhance and increase utilization of existing HIV and SRH services by reminding clients about safe sex methods available to them and providing a conduit for additional support.
  Interventions: Other: Automated text and voice messages
- Control Group (No Intervention): Those in the control group will get one "check-in" text or voice message between baseline and midline and another between midline and endline.

INTERVENTIONS:
Other: Automated text and voice messages — Participants will receive 3x weekly SMS or VM theory-based behavioral messages that will be designed to enhance and increase utilization of existing HIV and SRH services by reminding clients about safe sex methods available to them and providing a conduit for additional support. Participants will also be reminded in each message that they can talk to a peer counselor at any time by responding to the message. Participants who indicate they would like to talk to a counselor will receive a call from a Mobile Link community partner. The counselor will provide individualized information on HIV prevention and care and advice.
  Arms: Intervention Group

SUMMARY:
In Cambodia, HIV is prevalent in several high-risk groups including among female entertainment workers (FEWs) who work at entertainment venues such as karaoke bars and massage parlors and may engage in direct or indirect sex work. Reaching FEWs with sexual and reproductive health services such as testing and treatment for HIV and sexually transmitted infections (STIs) and contraception has been difficult because they are hidden and stigmatized. Mobile phone-based interventions may prove to be an effective way to reach this population and connect them with the existing services. This article describes study design and implementation of a two-arm randomized controlled trial of a mobile health intervention (the Mobile Link) aiming to improve sexual and reproductive health outcomes among FEWs in Cambodia. A two-armed randomized controlled trial (RCT) will be used to determine the effectiveness of a mobile phone-based text/voice messaging intervention. The intervention will be developed through a participatory process; 50 FEWs will work alongside researchers in focus groups to modify and tailor behavior change theory-based text and voice messages. Then, 600 FEWs will be recruited and randomly assigned into one of two arms: (1) a control group and (2) a mobile phone message group (either text messages or voice messages, delivery method chosen by participant). The primary outcome measures include HIV testing, condom use, STI testing and treatment and contraceptive use. If the Mobile Link trial is successful, an increase in condom use, screening and treatment for HIV and STI and contraception use is expected. These outcomes would lead to a reduction in the prevalence of HIV, STIs and unintended pregnancies. This trial is unique in a number of ways. First, the option of participation mode is offered to allow participants to choose the message medium that best links them to services. Second, this is the first RCT of a mobile phone-based behavior change intervention using SMS/VMs to support linkage to sexual and reproductive health services in Cambodia. Third, we are working with is a hidden, hard-to-reach and dynamic population with which traditional methods of outreach have not been fully successful.

DETAILED DESCRIPTION:
Introduction

Mobile phones are increasingly being used to enhance the effectiveness of health programs by engaging individuals in discreet and ongoing ways. Mobile phone health interventions, called mHealth, can also improve the availability and quality of operational research data. mHealth interventions have successfully been used in developing countries to collect health data, increase access to health knowledge and increase medication/appointment adherence. But, few mHealth interventions have been rigorously evaluated. There is strong evidence that mobile phone messages can be successfully used to support preventative healthcare, such as maternal postpartum visit attendance in Kenya. There is also evidence that self-report of risk behaviors through a mobile phone is a method of data collection that is as reliable and valid as in-person surveys. Especially for mobile or hidden populations in developing countries, mobile phones may become our most important tool for linking people to health services.

In Cambodia, several successful mobile phone-based health programs have been introduced in the areas of post-abortion contraceptive use, pharmacovigilence, diabetes self-management, case detection/notification and HIV education. The current evidence base for mobile phones used for health assessment and encouragement of the uptake of services, especially for hard-to-reach populations that face stigma and discrimination in developing countries is promising, but stronger impact evaluations are needed to understand the full benefits of such interventions.

One important hard-to-reach, high-risk group in Cambodia is the growing population of female entertainment workers (FEWs). FEWs are women working in entertainment venues such as karaoke bars, massage parlors, restaurants (as hostesses or singers) or beer gardens. FEWs frequently sell sex, directly or indirectly, to male patrons to supplement their income. By 2013, there were approximately 40,000 FEWs in Cambodia, 24,000 of whom resided in the capital city of Phnom Penh. This group has been increasing since the 2008 passage and implementation of the 'Law on Suppression of Human Trafficking and Sexual Exploitation,' which banned brothel-based sex work, and more women have moved into indirect sex work based out of entertainment venues.

The influx in the number of FEWs also follows the increase in garment factory jobs that attract young women from poor rural families to migrate to urban areas to earn and remit income to their families in their home villages. Today, the garment factories in Cambodia employ over 700,000 young women. Garment workers are typically not given fair wages, safe work environments or health insurance-a combination of factors that have resulted in worker unrests and mass fainting incidents at various factories. Claiming worker rights becomes a complicated challenge that involves risking their jobs, their livelihood and their ability to provide for family. As a result, more and more young migrant women become involved in alternative work opportunities in the entertainment industry. In addition, urban youth may also be at-risk of engaging in sex work. A recent study from Cambodia found that 48% of at-risk female youth across the country reported having been paid for sex in the past year.

FEWs in Cambodia are considered at high-risk for poor sexual and reproductive health (SRH) outcomes because of their involvement in direct or indirect sex work and limited access to SRH services. Recent studies indicate that HIV prevalence among women working in other entertainment establishments (9.8%), which is lower than street-based sex workers (37.3%) and brothel-based sex workers (17.4%), but is still considered a national concern. Recent data on HIV incidence among FEWs was 9.2% in 2009. In addition, incidences of C. trachomatis, Human papillomavirus and N. gonorrhea among FEWs are 11.5%, 41.1% and 7.8%, respectively.

Recent surveys on HIV testing rates indicate that 81.7% of FEWs reported ever having had an HIV test, and 52.3% reported having had an HIV test in the past six months. While there have been increases in reported condom use in commercial sex work over the past decade, there may be misreporting of condom use as well as condom failure. Consistent condom use is highly variable depending on the nature of relationship and several other factors. In 2014, our study of 667 FEWs showed that, in the past three months, 63.9% were able to find condoms when needed, and 38.2% used condoms at last sex with non-commercial partners. In another study, consistent condom use between FEWs and a native client was 98.8%. Consistent condom use among FEWs and non-commercial partners, such as boyfriends or other romantic relationships, in the past three months is estimated to be 26.5-34.1%, and has been reported to be as low as 20.6% among non-paying partners. Moreover, recent studies have shown that 21.4% of FEWs have had induced abortions since working in entertainment. Sexually transmitted infection (STI) diagnoses are also common among FEWs.

In Cambodia, government and Non-governmental organization providers currently offer free and widely available SRH services to FEWs. However, some FEWs experience barriers to using these services such as discrimination by providers. FEWs report a preference for private providers as a result. KHANA, the largest national HIV organization in Cambodia, is currently offering specialized services for FEWs including free distribution of condoms, a 'safe space' drop-in center, community-based finger-prick HIV and syphilis testing, accompanied referrals to enrolment of HIV-positive FEWs to pre-antiretroviral therapy (ART) and ART services, the integration of SRH services with HIV services, partner tracing and prevention of mother to child transmission (PMTCT) programming. Increasing utilization of these services by FEWs is a high priority.

The Mobile Link intervention is an operational mHealth research project that aims to engage FEWs, and link them to the existing high quality prevention, care and treatment services in the country. This intervention will consist of theory-based text, i.e. short message service (SMS), or voice messages (VM) that aim to increase the utilization of SRH services and reduce risk behaviors of FEWs in Cambodia. In addition, this intervention will determine if SMS/VM messaging can be a reliable source of monitoring and evaluation data. The initial operational research project will focus on FEWs as a proof of concept and if effective, the Mobile Link intervention program will be tailored for other key populations.

Cellphone use in Cambodia Cambodia is the first country in the world where the number of mobile phone users has surpassed the number of fixed landlines. The number of mobile subscribers in Cambodia reached 20 million at the end of 2013, surpassing the country's population by about 5 million. In a survey of 2,597 youth aged 15-24 drawn from all 24 provinces in Cambodia, 96% declared that they had access to a phone, with 68% reporting that they owned a personal mobile phone, and 72% had a mobile in their home. There are seven mobile phone service providers who continue to lower prices causing mobile phone use to become more affordable and penetration increases. Of the seven cellphone companies, SMART phone is the leader in overall number of subscribers, and Metphone has the most youth subscribers (68%).

The percentage of Cambodian people who own at least one smartphone, a cellular phone that performs many of the functions of a computer, typically having a touchscreen interface, Internet access, and an operating system capable of running downloaded applications, was 39.5% in 2015, almost doubling the 2013 figure. Controlling for location and gender, 51.3% of people between the ages of 15 and 65 in 2015 had at least one phone through which it was possible to send and receive messages in Khmer script (a 65% increase from last year). The growth in the use of phones that can text Khmer script for women in the last year was 89.8%; while for men it was only 61.8%. The ability to display Khmer was also found to gradually increase with the level of education of the owner, from 33% of those who had no formal education to 69.2% for those who attended or have completed university.

In a recent report from the United Nations Development Program (UNDP), of 2,597 Cambodian people between the ages of 15-24, 98% reported that they used their mobile phones mostly for making and receiving calls, 43% for listening to the radio and 32% for sending and receiving messages, followed relatively closely by playing and downloading games (27%) and taking photos (22%). Of those youth who used SMS, the majority used English language messages (81%). In the Asian-Pacific countries, the number of mobile social media users was set to reach one billion by the fourth quarter of 2015; and in Cambodia increasing 108% from the previous year. The number of people in the region accessing social media from mobile devices jumped an impressive 32% in the past year, to reach 900 million. In Cambodia, about 80% of the traffic is driven by Facebook and YouTube. The proliferation of smartphones has catapulted Facebook to Cambodia's second-most important source of news this year, surpassing radio and edging ever closer to overtaking television.

Entertainment workers have both smart and basic mobile phones, use them daily to text and engage in social media and have expressed interest in receiving health information through their phones.

Objectives The overall goal of the study is to deploy and rigorously evaluate the efficacy of Mobile Link, an innovative intervention to engage young FEWs in Cambodia through frequent SMS/VMs that link them to existing high-quality services including HIV testing. A 12-month randomized controlled trial (RCT) will be conducted to evaluate the Mobile Link intervention, with two arms of 300 FEWs each. FEWs will be equally randomized into one of two groups: (1) no intervention and (2) SMS or VM theory-based behavioral messages.

Specific objectives include: (1) developing the Mobile Link intervention for young FEWs in Cambodia by conducting participant observation, focus groups and cognitive pilot interviews to produce a bank of 600 theory-informed SMS/VM messages as well as pilot testing the feasibility of collecting data from FEWs through SMS and VMs; 2) evaluating the efficacy of the Mobile Link intervention at the individual and venue level for increasing the uptake of HIV testing, condom use and the utilization of comprehensive SRH care services among 600 sexually-active FEWs through a 12 month, 2-armed RCT and (3) determining the cost-effectiveness of the Mobile Link intervention for FEWs as compared the standard outreach, care and treatment services provided by KHANA.

ELIGIBILITY:
Inclusion Criteria:

All participants must:

* live and work at an entertainment venue in Cambodia;
* currently sexually active defined as engaged in oral, vaginal or anal sex in the past 3 months;
* own their own mobile phone;
* know how to retrieve VM or retrieve and read SMS on mobile phone (Khmer or Khmer with English alphabet);
* self-identify as a FEW;
* are willing to receive at most one SMS/VM per day for one year;
* provide written informed consent and
* agree to a follow-up visit after six months and 12 months.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — They must be biologically female.
Enrollment: 600 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Recent HIV Testing | past 6 months
  Having had an HIV test in the past 6 months
Condom Use with Clients | Past 1 month
  Frequency of Condom Use with Clients in past month (always, sometime, rarely, never)
Condom Use with boyfriend/husband/romantic partner | Past 1 month
  Frequency of Condom Use with boyfriend/husband/romantic partner in past month (always, sometime, rarely, never)
Contraceptive Prevalence Rate | Past 1 month
  Currently using modern Contraceptive method if trying to prevent pregnancy
Abortion Rate | Past 6 months
  Abortion in last six months
Workplace Alcohol Consumption | Past 6 months
  Forced alcohol consumption at work in past six months
Gender-Based harassment rate | Past 6 months
  Experienced unwanted touching or groping in the past six months
Gender-based violence rate | Past 6 months
  Has experienced verbal abuse such as threats of violence, physical violence, rape/sexual assault in the past six months
STI Screening | Past six months
  Sought treatment when experiencing STI symptoms in past 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- KHANA, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gisore P, Shipala E, Otieno K, Rono B, Marete I, Tenge C, Mabeya H, Bucher S, Moore J, Liechty E, Esamai F. Community based weighing of newborns and use of mobile phones by village elders in rural settings in Kenya: a decentralised approach to health care provision. BMC Pregnancy Childbirth. 2012 Mar 19;12:15. doi: 10.1186/1471-2393-12-15. PMID 22429731
- [Background] Curran K, Mugo NR, Kurth A, Ngure K, Heffron R, Donnell D, Celum C, Baeten JM. Daily short message service surveys to measure sexual behavior and pre-exposure prophylaxis use among Kenyan men and women. AIDS Behav. 2013 Nov;17(9):2977-85. doi: 10.1007/s10461-013-0510-4. PMID 23695519
- [Background] Hossain M, Mani KK, Sidik SM, Hayati KS, Rahman AK. Randomized controlled trial on drowning prevention for parents with children aged below five years in Bangladesh: a study protocol. BMC Public Health. 2015 May 11;15:484. doi: 10.1186/s12889-015-1823-1. PMID 25957574
- [Background] Crawford J, Larsen-Cooper E, Jezman Z, Cunningham SC, Bancroft E. SMS versus voice messaging to deliver MNCH communication in rural Malawi: assessment of delivery success and user experience. Glob Health Sci Pract. 2014 Jan 28;2(1):35-46. doi: 10.9745/GHSP-D-13-00155. eCollection 2014 Feb. PMID 25276561
- [Background] Dammert AC, Galdo JC, Galdo V. Preventing dengue through mobile phones: evidence from a field experiment in Peru. J Health Econ. 2014 May;35:147-61. doi: 10.1016/j.jhealeco.2014.02.002. Epub 2014 Mar 5. PMID 24681813
- [Background] Free C, Phillips G, Galli L, Watson L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technology-based health behaviour change or disease management interventions for health care consumers: a systematic review. PLoS Med. 2013;10(1):e1001362. doi: 10.1371/journal.pmed.1001362. Epub 2013 Jan 15. PMID 23349621
- [Background] Deglise C, Suggs LS, Odermatt P. SMS for disease control in developing countries: a systematic review of mobile health applications. J Telemed Telecare. 2012 Jul;18(5):273-81. doi: 10.1258/jtt.2012.110810. Epub 2012 Jul 23. PMID 22826375
- [Background] Mushamiri I, Luo C, Iiams-Hauser C, Ben Amor Y. Evaluation of the impact of a mobile health system on adherence to antenatal and postnatal care and prevention of mother-to-child transmission of HIV programs in Kenya. BMC Public Health. 2015 Feb 7;15:102. doi: 10.1186/s12889-015-1358-5. PMID 25886279
- [Background] Raifman JR, Lanthorn HE, Rokicki S, Fink G. The impact of text message reminders on adherence to antimalarial treatment in northern Ghana: a randomized trial. PLoS One. 2014 Oct 28;9(10):e109032. doi: 10.1371/journal.pone.0109032. eCollection 2014. PMID 25350546
- [Background] Sabin LL, Bachman DeSilva M, Gill CJ, Zhong L, Vian T, Xie W, Cheng F, Xu K, Lan G, Haberer JE, Bangsberg DR, Li Y, Lu H, Gifford AL. Improving Adherence to Antiretroviral Therapy With Triggered Real-time Text Message Reminders: The China Adherence Through Technology Study. J Acquir Immune Defic Syndr. 2015 Aug 15;69(5):551-9. doi: 10.1097/QAI.0000000000000651. PMID 25886927
- [Background] Islam SM, Lechner A, Ferrari U, Froeschl G, Alam DS, Holle R, Seissler J, Niessen LW. Mobile phone intervention for increasing adherence to treatment for type 2 diabetes in an urban area of Bangladesh: protocol for a randomized controlled trial. BMC Health Serv Res. 2014 Nov 26;14:586. doi: 10.1186/s12913-014-0586-1. PMID 25424425
- [Background] Vodopivec-Jamsek V, de Jongh T, Gurol-Urganci I, Atun R, Car J. Mobile phone messaging for preventive health care. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD007457. doi: 10.1002/14651858.CD007457.pub2. PMID 23235643
- [Background] Esbensen BA, Thomsen T, Hetland ML, Beyer N, Midtgaard J, Loppenthin K, Jennum P, Ostergaard M, Sorensen J, Christensen R, Aadahl M. The efficacy of motivational counseling and SMS-reminders on daily sitting time in patients with rheumatoid arthritis: protocol for a randomized controlled trial. Trials. 2015 Jan 27;16:23. doi: 10.1186/s13063-014-0540-x. PMID 25623388
- [Background] Youl PH, Soyer HP, Baade PD, Marshall AL, Finch L, Janda M. Can skin cancer prevention and early detection be improved via mobile phone text messaging? A randomised, attention control trial. Prev Med. 2015 Feb;71:50-6. doi: 10.1016/j.ypmed.2014.12.009. Epub 2014 Dec 16. PMID 25524612
- [Background] Smith C, Vannak U, Sokhey L, Ngo TD, Gold J, Free C. Mobile Technology for Improved Family Planning (MOTIF): the development of a mobile phone-based (mHealth) intervention to support post-abortion family planning (PAFP) in Cambodia. Reprod Health. 2016 Jan 5;13:1. doi: 10.1186/s12978-015-0112-x. PMID 26728505
- [Background] Odeny TA, Bukusi EA, Cohen CR, Yuhas K, Camlin CS, McClelland RS. Texting improves testing: a randomized trial of two-way SMS to increase postpartum prevention of mother-to-child transmission retention and infant HIV testing. AIDS. 2014 Sep 24;28(15):2307-12. doi: 10.1097/QAD.0000000000000409. PMID 25313586
- [Background] Swendeman D, Comulada WS, Ramanathan N, Lazar M, Estrin D. Reliability and validity of daily self-monitoring by smartphone application for health-related quality-of-life, antiretroviral adherence, substance use, and sexual behaviors among people living with HIV. AIDS Behav. 2015 Feb;19(2):330-40. doi: 10.1007/s10461-014-0923-8. PMID 25331266
- [Background] Swendeman D. Are mobile phones the key to HIV prevention for mobile populations in India? Indian J Med Res. 2013 Jun;137(6):1024-6. No abstract available. PMID 23852282
- [Background] Smith C, Vannak U, Sokhey L, Ngo TD, Gold J, Khut K, Edwards P, Rathavy T, Free C. MObile Technology for Improved Family Planning Services (MOTIF): study protocol for a randomised controlled trial. Trials. 2013 Dec 12;14:427. doi: 10.1186/1745-6215-14-427. PMID 24330763
- [Background] Baron S, Goutard F, Nguon K, Tarantola A. Use of a text message-based pharmacovigilance tool in Cambodia: pilot study. J Med Internet Res. 2013 Apr 16;15(4):e68. doi: 10.2196/jmir.2477. PMID 23591700
- [Background] van Olmen J, Ku GM, van Pelt M, Kalobu JC, Hen H, Darras C, Van Acker K, Villaraza B, Schellevis F, Kegels G. The effectiveness of text messages support for diabetes self-management: protocol of the TEXT4DSM study in the democratic Republic of Congo, Cambodia and the Philippines. BMC Public Health. 2013 May 1;13:423. doi: 10.1186/1471-2458-13-423. PMID 23635331
- [Background] Lorent N, Choun K, Thai S, Kim T, Huy S, Pe R, van Griensven J, Buyze J, Colebunders R, Rigouts L, Lynen L. Community-based active tuberculosis case finding in poor urban settlements of Phnom Penh, Cambodia: a feasible and effective strategy. PLoS One. 2014 Mar 27;9(3):e92754. doi: 10.1371/journal.pone.0092754. eCollection 2014. PMID 24675985
- [Background] Brody C, Chhoun P, Tuot S, Pal K, Chhim K, Yi S. HIV risk and psychological distress among female entertainment workers in Cambodia: a cross-sectional study. BMC Public Health. 2016 Feb 9;16:133. doi: 10.1186/s12889-016-2814-6. PMID 26861542
- [Background] Brody C, Tuot S, Chhea C, Saphonn V, Yi S. Factors associated with sex work among at-risk female youth in Cambodia: a cross-sectional study. AIDS Care. 2016;28(3):339-46. doi: 10.1080/09540121.2015.1096893. Epub 2015 Oct 19. PMID 26477781
- [Background] Yi S, Tuot S, Chhoun P, Pal K, Tith K, Brody C. Factors associated with induced abortion among female entertainment workers: a cross-sectional study in Cambodia. BMJ Open. 2015 Jul 31;5(7):e007947. doi: 10.1136/bmjopen-2015-007947. PMID 26231754
- [Background] Page K, Stein E, Sansothy N, Evans J, Couture MC, Sichan K, Cockroft M, Mooney-Somers J, Phlong P, Kaldor J, Maher L; Young Women's Health Study Collaborative*. Sex work and HIV in Cambodia: trajectories of risk and disease in two cohorts of high-risk young women in Phnom Penh, Cambodia. BMJ Open. 2013 Sep 10;3(9):e003095. doi: 10.1136/bmjopen-2013-003095. PMID 24022389
- [Background] Couture MC, Sansothy N, Sapphon V, Phal S, Sichan K, Stein E, Evans J, Maher L, Kaldor J, Vun MC, Page K. Young women engaged in sex work in Phnom Penh, Cambodia, have high incidence of HIV and sexually transmitted infections, and amphetamine-type stimulant use: new challenges to HIV prevention and risk. Sex Transm Dis. 2011 Jan;38(1):33-9. doi: 10.1097/OLQ.0b013e3182000e47. PMID 21085056
- [Background] Couture MC, Page K, Stein ES, Sansothy N, Sichan K, Kaldor J, Evans JL, Maher L, Palefsky J. Cervical human papillomavirus infection among young women engaged in sex work in Phnom Penh, Cambodia: prevalence, genotypes, risk factors and association with HIV infection. BMC Infect Dis. 2012 Jul 28;12:166. doi: 10.1186/1471-2334-12-166. PMID 22839728
- [Background] Yi S, Tuot S, Chhoun P, Brody C, Tith K, Oum S. The impact of a community-based HIV and sexual reproductive health program on sexual and healthcare-seeking behaviors of female entertainment workers in Cambodia. BMC Infect Dis. 2015 Jun 6;15:221. doi: 10.1186/s12879-015-0954-4. PMID 26047818
- [Background] Maher L, Mooney-Somers J, Phlong P, Couture MC, Kien SP, Stein E, Bates AJ, Sansothy N, Page K; Young Women's Health Study Collaborative. Condom negotiation across different relationship types by young women engaged in sex work in Phnom Penh, Cambodia. Glob Public Health. 2013;8(3):270-83. doi: 10.1080/17441692.2013.767930. Epub 2013 Feb 22. PMID 23432108
- [Background] Bui TC, Markham CM, Tran LT, Beasley RP, Ross MW. Condom negotiation and use among female sex workers in Phnom Penh, Cambodia. AIDS Behav. 2013 Feb;17(2):612-22. doi: 10.1007/s10461-012-0369-9. PMID 23196858
- [Background] Brody C, Tatomir B, Sovannary T, Pal K, Mengsrun S, Dionosio J, Luong MA, Yi S. Mobile phone use among female entertainment workers in Cambodia: an observation study. Mhealth. 2017 Jan 30;3:3. doi: 10.21037/mhealth.2017.01.01. eCollection 2017. PMID 28293620
- [Derived] Avancena ALV, Brody C, Chhoun P, Tuot S, Yi S. Connecting Female Entertainment Workers in Cambodia to Health Care Services Using mHealth: Economic Evaluation of Mobile Link. JMIR Form Res. 2024 Jul 25;8:e52734. doi: 10.2196/52734. PMID 39052328
- [Derived] Brody C, Chhoun P, Tuot S, Fehrenbacher AE, Moran A, Swendeman D, Yi S. A Mobile Intervention to Link Young Female Entertainment Workers in Cambodia to Health and Gender-Based Violence Services: Randomized Controlled Trial. J Med Internet Res. 2022 Jan 4;24(1):e27696. doi: 10.2196/27696. PMID 34982716
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Brody C, Tuot S, Chhoun P, Swendeman D, Kaplan KC, Yi S. Mobile Link - a theory-based messaging intervention for improving sexual and reproductive health of female entertainment workers in Cambodia: study protocol of a randomized controlled trial. Trials. 2018 Apr 19;19(1):235. doi: 10.1186/s13063-018-2614-7. PMID 29673381